CLINICAL TRIAL: NCT00203632
Title: A Trial of the Effect of Rosiglitazone as Add on to Metformin Therapy on Endothelial Function in Subjects With Type II DM
Brief Title: Glitazones and Endothelial Function (GATE)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated at 50% enrollment due to recent concerns about rosiglitazone
Sponsor: University of Calgary (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPD 084385
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; endothelium; thiazolidinediones; atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rosiglitazone/placebo

SUMMARY:
The purpose of the study is to determine if the addition of rosiglitazone to subjects with fair glucose control on other oral agents improves endothelial function, a surrogate marker of vascular health.

It is hypothesized that improving whole body insulin sensitivity with combination therapy including rosiglitazone will restore the vascular actions of insulin and improve endothelium-dependent vasomotion more effectively than placebo in patients with diabetes mellitus.

DETAILED DESCRIPTION:
The vascular endothelium has emerged as a critical determinant of cardiovascular health and disease, and improving endothelial function is an important target for therapy. Accumulating evidence suggest that insulin resistance in patients with diabetes and the metabolic syndrome may impair endothelial function, uncovering a proinflammatory, and proatherosclerotic vascular phenotype. The GATE study (Glitazones And The Endothelium) is a randomized, double blind study to evaluate the effects of rosiglitazone vs. placebo on endothelial function when employed as an add-on therapy in diabetic patients currently treated with oral therapy. We hypothesize that the PPAR-gamma agonist rosiglitazone, will improve endothelium-dependent vasodilatation, and that this effect will be related to improvements in insulin sensitivity, with concomitant reductions in whole body insulin resistance. Furthermore, the beneficial effects of rosiglitazone will be additive to existing oral therapies that may modulate endothelial function, such as metformin. Since endothelial dysfunction plays a pivotal role in the development and progression of atherosclerosis, these studies may provide the rationale and impetus for aggressive treatment of insulin resistant patients with glitazone therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients (both men and women) considered for participation in GATE study have to be non-insulin dependent diabetics (according to Canadian Diabetes Association criteria, namely a fasting serum glucose ≥ 7.0 mmol/L on two occasions, a casual glucose ≥ 11.1 mmol/l with symptoms, or a 2-h post-oral glucose tolerance test glucose of ≥ 11.1 mmol/l) with unsatisfactory glycemic control on oral therapy (HbA1c 6-10%).

Exclusion Criteria:

* Exclusion criteria includes, congestive heart failure (NYHA class III & IV or ejection fraction less than 35%), poorly controlled hypertension (blood pressure > 160/90), hypercholesterolemia (total cholesterol > 6.2 mmol/l), hypertriglyceridemia (triglycerides > 4.0 mmol/l), poor or excellent control of DM (HgA1c <6 % or HbA1c > 10% respectively), known diabetic retinopathy, age at diagnosis of diabetes less than 25 years, current participation in another clinical trial and contraindications to glitazones therapy, including renal (creatinine > 200 micromol/ L) or hepatic (ALT > 2.5 times the upper limit of normal) impairment and/ or known intolerance to glitazones. Patients must be stable on medications that affect endothelial function for more than one month. This includes ACE-inhibitors, angiotensin receptor blockers, statins, calcium channel blockers, hormone replacement therapy and anti-oxidant vitamins, including folates. Patients on insulin will be excluded. Patients in whom it is felt that attainment of better glucose control is required within 3 months will also be excluded. Patients with stable coronary disease will be eligible for the study as long as they are > one month post myocardial infarction, percutaneous intervention or bypass surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary end-point of the study is the percent change in forearm blood flow to acetylcholine in patients randomized to rosiglitazone compared with placebo.

SECONDARY OUTCOMES:
Secondary end-points include (i) the percent change in forearm blood flow to verapamil and the absolute change to both acetylcholine and verapamil and (ii) the relationship between HOMA-IR, CRP and endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Todd J Anderson, MD, Principal Investigator — University of Calgary; Subodh Verma, MD, PhD, Study Chair — University of Toronto
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Hubacek J, Verma S, Shewchuk L, Ross SJ, Edwards A, Anderson TJ. Rationale and design of the Glitazones and the Endothelium (GATE) study: evaluation of rosiglitazone on endothelial function in patients with diabetes. Can J Cardiol. 2004 Dec;20(14):1449-53. PMID 15614340